CLINICAL TRIAL: NCT07348458
Title: The Effect of Intraoperative Thermal Kidney Insulation on Current Kidney Transplantation Surgical Practices
Brief Title: Kidney Protective Jacket
Acronym: KPJ
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: iiShield (Industry)
Collaborators: Western Sydney Local Health District (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: CI-TPL-01
Record Dates: First submitted 2025-12-18; First posted 2026-01-16 (Actual); Last update posted 2026-01-16 (Actual); Status verified 2026-01

CONDITIONS: Kidney Transplant
Keywords: Kidney transplant; Renal transplant; Second warm ischaemic time; Ischaemia-reperfusion injury; Kidney Protective Jacket; Graft cooling
MeSH Terms: conditions — Reperfusion Injury

STUDY DESIGN:
Masking Description: Participant and outcomes assessor will be blinded
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- Kidney Protective Jacket (Experimental): Application of the KPJ to the renal transplant.
  Interventions: Device: Kidney Protective Jacket

INTERVENTIONS:
Device: Kidney Protective Jacket — The KPJ™ is a novel thermal insulating protective jacket specifically designed to be applied to the kidney during transplant anastomoses, or the SWIT interval. It is applied prior to removing the kidney from cold storage, and remains on for the duration of anastomoses, after which it can be easily removed.
  The Kidney Protective Jacket (KPJ) was designed and developed in accordance with ISO 13485 and 21 CFR 820 design control requirements. Throughout the development process, relevant standards were applied, including those related to risk management (ISO 14971), usability engineering (IEC 62366), biocompatibility of materials (ISO 10993 series), and sterilisation validation (ISO 11137).
  Manufacturing is carried out by an ISO 13485-certified contract manufacturer, with processes including injection moulding of medical-grade silicone, assembly of the sterile barrier system (comprising a medical-grade plastic tray and Tyvek® seal), and final device packaging. Sterilisation is performed us

SUMMARY:
This is a safety study designed to investigate the safety of utilizing the Kidney Protective Jacket (KPJ)™ during kidney transplantation. In general, we aim to use the device in all possible recipients, aiming to demonstrate its safety in the variable circumstances that may arise during kidney transplantation, e.g. single or multiple renal vessels, different-sized kidneys, and variable recipient size and weight.

DETAILED DESCRIPTION:
Kidneys obtained from organ donors necessarily undergo a period of ischemia whereby there is no blood supply or oxygenation of the kidney until the kidney is implanted into the transplant recipient. During organ retrieval, the kidney is flushed with cold preservation fluid, after which it is most commonly placed in cold storage (CS) solution until the kidney is implanted. This method reliably keeps the kidney cool, dropping its metabolic rate and ATP consumption, and aiming to minimize the ischemia-reperfusion injury (IRI) which is one of key determinants of early and longer-term graft outcomes (1).

However, once the kidney is ready for transplantation, it must be removed from CS in preparation for anastomoses in the recipient. The kidney at this stage is exposed to the 37°C environment of the patient's body temperature and begins to re-warm; this interval is known as the second warm ischemic time (SWIT). After it reaches a temperature of 15°C to 18°C, the degree of renal glomerular and tubular metabolic activity results in warm ischemic damage (2-5). The SWIT usually ranges between 15-70 minutes, depending on the number of vessels to be reattached, surgeon experience, and anatomical differences (6-10).

Multiple studies have demonstrated the changes that occur in kidney temperature during the transplantation process. A study by Feuillu et al. (2003) on 65 patients showed that mean kidney temperature at the time of removal from the cold storage was 1.6°C and 6.3°C when the kidney was placed in the recipient (3). Then, kidney temperature increased logarithmically reaching mean kidney temperature of 26.7°C at end of anastomosis (mean SWIT: 45.5 [22-85] min). Kidney warming speed was 0.48°C/min and was dependent on the length of time of vascular anastomosis (3). The other series on 152 consecutive adult living donor kidney transplantations showed the mean SWIT was 41.3 ± 10.1 minutes with a temperature of 5.4 °C at baseline which gradually increased to 13.7, 17.4, and 20.2°C after 10, 20, and 30 min, respectively (4). The percentage of kidneys with a temperature of 15°C or higher was 81.2% after 20 min and 97.5% after 30 min (4).

There is large scale registry data that demonstrates the deleterious impact of kidney rewarming during the SWIT on subsequent transplant outcomes. In particular, using large cohorts from Europe, Heylen et al demonstrated: (i) increased risk with respect to higher rates of delayed graft function (defined as the need for dialysis in the 1st week post transplant), quantified as an odds ratio of 1.05 for every additional minute (i.e. 5% additional risk for every minute); (ii) poorer kidney transplant function up to 3 years post-transplant; and (iii) elevated rates of death-censored graft failure (hazard ratio of 1.10) for every additional 10 minutes. This includes outcomes for all types of deceased donor kidneys (8). The longer the SWIT the worse the outcome - this effect is especially pronounced in circulatory death donors.

Maintenance of appropriate renal hypothermia is, therefore, not only important during preservation and transportation, but also when the kidney is removed from its cooled transport media in preparation for anastomoses (8,10). This cannot be achieved using current core cooling methods (i.e. direct intravascular perfusion) during anastomoses but must rely upon external methods and/or devices. Various examples of such devices and/or techniques exist, although they have had limited success, limited generalizability, impede surgical vision, and are prone to inconsistencies. There is currently no commercial product that allows cooling of the kidney to minimise the impacts of the SWIT time.

With this current context, we wish to undertake a trial of a novel device, the Kidney Protective Jacket (KPJ™), which will assess its usability and establish its safety in the clinical setting, and add significantly to worldwide knowledge of this process. Ultimately, this device aims to provide consistent user experience with good thermoregulation leading to minimisation of IRI from the SWIT. We anticipate this will translate into improving the recipient's transplant outcomes.

ELIGIBILITY:
Inclusion Criteria:

* All deceased and living donor kidneys that are deemed suitable for transplantation
* All suitable recipients who are 18 years or greater, and undergoing their first or second kidney transplant
* All recipients must be able to provide full informed consent

Exclusion Criteria:

* Paediatric donor kidneys (kidneys from donors < 16 years in age)
* Patients with a known allergy or hypersensitivity to silicone

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Estimated)
Dates: Start 2026-01-01 (Estimated); Primary Completion 2026-06-30 (Estimated); Study Completion 2026-12-31 (Estimated)

PRIMARY OUTCOMES:
Safety of the Kidney Protective Jacket | Until 20 participants are recruited, baseline participant characteristics collected pre-operatively, intra-operative times noted, and incidence of serious adverse events at 30 days post procedure.
  The primary objective is to assess the safety of use of KPJ™ (per its intended use) during kidney transplantation. Specifically, we are assessing the proportion of participants sustaining Serious Adverse Effects directly attributable to KPJ use (i.e., Serious Adverse Device Events [SADE]) in the time period of 30 days post transplantation. We also want to examine the safety in variable circumstances, e.g. single and multiple renal vessels, different sized kidneys, variable recipient size and weights.

SECONDARY OUTCOMES:
Device related events | When 20 participants have been recruited and 30 days post transplantation procedure.
  Non-serious adverse device effects (n) and Non-device-related adverse events (n)
Temperature change during SWIT (°C) | When 20 participants have been recruited and 30 days post transplantation procedure.
  Temperature change during SWIT (°C)
Surgery time (minutes) | When 20 participants have been recruited and 30 days post transplantation procedure.
  Surgery time (minutes)
Delayed graft function (%) | When 20 participants have been recruited and 30 days post transplantation procedure.
  Delayed graft function (%)
Serum creatinine (μmol/L) | When 20 participants have been recruited and 30 days post transplantation procedure.
  Serum creatinine (μmol/L)
Estimated glomerular filtration rate - eGFR (mL/min) | When 20 participants have been recruited and 30 days post transplantation procedure.
  Estimated glomerular filtration rate - eGFR (mL/min)
Graft survival | 30 days post transplantation procedure.
  At 30 days post procedure - yes or no answer to the question

IPD SHARING:
Plan to Share IPD: No
The other investigators will be informed once this application is approved, however will not need to review it / have it shared